CLINICAL TRIAL: NCT01394198
Title: Correlation of Somatic Dysfunction With Gastrointestinal Endoscopic Findings
Status: Completed | Type: Observational
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 101123-001
Record Dates: First submitted 2011-06-27; First posted 2011-07-14 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Segmental and Somatic Dysfunction; Pathological Conditions, Signs and Symptoms; Ectopic Intestinal Mucosa
Keywords: Osteopathic Manipulative Medicine (OMM); Neuromuscular Medicine (NMM); Somatic Dysfunction; Correlational Study; Endoscopy
MeSH Terms: conditions — Pathological Conditions, Signs and Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to correlate the link between palpatory findings of somatic dysfunction and gastrointestinal endoscopic evidence of changes in mucosa. The investigators' hypothesis is that there is a direct connection between somatic palpatory changes and intestinal mucosal changes via a somatovisceral/viscerosomatic mechanism.

DETAILED DESCRIPTION:
The study protocol is limited to an extra physical examination (the focused structural exam) prior to a scheduled routine or diagnostic endoscopy. Immediately prior to the scheduled endoscopy, subjects enrolled in the study will be palpated by a Neuromuscular Medicine (NMM)/Osteopathic Manipulative Medicine (OMM) specialist for spinal tenderness, tissue texture changes and asymmetry or restricted range of motion as well as tenderness of Chapman points. The entire spine from the occipitoatlantal joint to the sacrum will be evaluated along with specific intercostal abdominal and lower extremity areas. The positive structural examination findings of spinal tenderness, tissue texture changes and asymmetry or restricted range of motion will be compared to the visual and pathological findings recorded in the operative report of the endoscopy procedure and the pathological report of any biopsies obtained during the endoscopic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients already scheduled for upper or lower endoscopy at Kirksville Family Medicine Clinic
* Must be 21 years of age or older
* Subjects must be able to lie in the prone position for 30 minutes

Exclusion Criteria:

* Subjects cannot have history of spinal fractures or surgical intervention of the spine that could alter the palpatory findings of the spinal and paraspinal regions
* Subjects who are wards of the state or are unable to sign the consent form on their own behalf will be excluded
* Subjects will be excluded if they are unable to lie prone for 30 minutes
* Subjects will be excluded if they are not already scheduled for an endoscopy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 21 years of age or older, of the Kirksville College of Osteopathic Family Medicine Clinic, and are scheduled for upper or lower endoscopy based on clinical symptomology or for routine screening based on age or risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Osteopathic structural exam findings of somatic dysfunction | Structural exam will be conducted prior to the scheduled endoscopy on the same day. The results will be recorded on a somatic dysfunction findings worksheet during the exam. This exam will only occur one time on the day of the endoscopy.
  A musculoskeletal exam will be done by a Neuromuscular Medicine (NMM)/Osteopathic Manipulative Medicine (OMM) specialist for spinal tenderness, tissue texture changes, asymmetry, and restricted range of motion as well as tenderness of Chapman Points. The entire spine from the occipitoatlantal joint to the sacrum will be evaluated along with specific intercostal abdominal and lower extremity areas. The exam will identify whether tenderness, tissue texture changes, asymmetry, and range of motion restrictions exist at each of the vertebral segments.

CONTACTS AND LOCATIONS:
Overall Officials: Karen T Snider, D.O., Principal Investigator — Kirksville College of Osteopathic Medicine; AT Still University
Locations (1):
- Kirksville College of Osteopathic Medicine Family Practice Clinic, Kirksville, Missouri, United States

REFERENCES:
- [Derived] Snider KT, Schneider RP, Snider EJ, Danto JB, Lehnardt CW, Ngo CS, Johnson JC, Sheneman TA. Correlation of Somatic Dysfunction With Gastrointestinal Endoscopic Findings: An Observational Study. J Am Osteopath Assoc. 2016 Jun 1;116(6):358-69. doi: 10.7556/jaoa.2016.076. PMID 27214772